CLINICAL TRIAL: NCT03303235
Title: How's the Tone? Intravenous Versus Intramuscular Administration of Methylergonovine for Uterine Contraction in Cesarean Sections
Brief Title: Intravenous Versus Intramuscular Administration of Methylergonovine for Uterine Contraction in Cesarean Sections
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Collaborators left the institution.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00120873
Record Dates: First submitted 2017-09-26; First posted 2017-10-05 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Uterine Atony; Uterine Tone Disorders; Postpartum Hemorrhage
Keywords: methylergonovine
MeSH Terms: conditions — Uterine Inertia; Postpartum Hemorrhage | interventions — Methylergonovine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient and obstetrician will all be blinded to group assignments. The anesthesiologist will make and administer the medication, as it is important for timely administration of the methylergonovine when it is asked to be used. The anesthesiologist directly taking care of the patient will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IV Methergine (Experimental): IV methylergonovine group
  -IM 0.9% NaCl (1 ml)) + IV methylergonovine (2 mcg/ml) infusion (100 ml)
  Interventions: Drug: Methylergonovine
- Conventional (Active Comparator): IM methylergonovine group
  -200 mcg IM methylergonovine (1 ml) + IV 0.9% NaCl infusion (100 ml)
  Interventions: Drug: Methylergonovine

INTERVENTIONS:
Drug: Methylergonovine — IV vs IM
  Other Names: methergine

SUMMARY:
Insufficient uterine tone resulting in atony can potentiate hemorrhage and adverse outcomes for the parturient. Oxytocin is the first pharmacologic agent used, followed by methylergonovine, carboprost, and misoprostol. The American Congress of Obstetricians and Gynecologists (ACOG) recommends the sequential use of oxytocin, followed by methylergonovine, carboprost, misoprostol, then surgical intervention for cases of refractory uterine atony. Many studies have examined the effect and dosage of intravenous uterotonics, including oxytocin.

Although there are anecdotal reports of using intravenous bolus or rapid infusion of methylergonovine, no randomized trial has compared efficacy and side effects of these two routes of administration. Investigators hypothesize that intravenous methylergonovine reduces the time to adequate uterine tone (the tone at which the uterus is adequately contracted to prevent atony after delivery of neonate), decreases the total dose of methylergonovine to contract the uterus, and therefore produces fewer side effects of hypertension, nausea, and vomiting. Reducing the time to achieve adequate uterine tone is likely to decrease postpartum hemorrhage.

DETAILED DESCRIPTION:
The United States is one of the few modern countries in which maternal peripartum mortality continues to rise. One of the three most important causes of maternal mortality is severe hemorrhage. Controlling postpartum uterine tone remains an important role for the obstetric anesthesiologist. Insufficient uterine tone resulting in atony can potentiate hemorrhage and adverse outcomes for the parturient. Oxytocin is the first pharmacologic agent used, followed by methylergonovine, carboprost, and misoprostol. The American Congress of Obstetricians and Gynecologists (ACOG) recommends the sequential use of oxytocin, followed by methylergonovine, carboprost, misoprostol, then surgical intervention for cases of refractory uterine atony. Many studies have examined the effect and dosage of intravenous uterotonics, including oxytocin.

Methylergonovine maleate is a semi-synthetic ergot alkaloid. Methylergonovine(200 mcg) is administered intramuscularly when oxytocin has been administered but has not contracted the uterus sufficiently. It is not without side effects, however. Due to its vasoconstrictive properties, methylergonovine has been shown to elevate blood pressures and is avoided in preeclamptic patients who may not tolerate abrupt increases in blood pressures. Although there are anecdotal reports of using intravenous bolus or rapid infusion of methylergonovine, no randomized trial has compared efficacy and side effects of these two routes of administration. Investigators hypothesize that intravenous methylergonovine reduces the time to adequate uterine tone (the tone at which the uterus is adequately contracted to prevent atony after delivery of neonate), decreases the total dose of methylergonovine to contract the uterus, and therefore produces fewer side effects of hypertension, nausea, and vomiting. Reducing the time to achieve adequate uterine tone is likely to decrease postpartum hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted for elective cesarean section
* All laboring patients for planned vaginal delivery as these women may have an unplanned cesarean delivery for maternal or for fetal indications
* Patients not in labor but admitted for non-elective cesarean section
* Administration of oxytocin prior to administration of methylergonovine, in accordance to the ACOG guideline for postpartum hemorrhage
* Obstetrician's request for methylergonovine intraoperatively to the anesthesiologist

Exclusion Criteria:

* Fetus not considered to be of viable gestational age by obstetrical team
* Patients with hypertension (either chronic or pregnancy-induced, including preeclampsia)
* Patients with coronary artery disease, established and diagnosed by medical internist or cardiologist
* Patients taking CYP3A4 inhibitors
* Patients taking beta blockers.
* Patients with contraindications to any of the uterotonic agents for whatever medical reason (allergies, for example)
* Surgeon request for administration of methylergonovine earlier than per protocol due to clinical situation as abovementioned
* Maternal or obstetrician refusal
* Patients who require obstetrical intervention before 30 minutes has elapsed

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female parturients eligible to undergo a cesarean section
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Time to achieve "adequate" uterine tone | 10 minutes
  Our primary objective is to determine the time to achieve "adequate" uterine tone with either intramuscular (IM) dose versus intravenous (IV) dose methylergonovine, when oxytocin has failed to do so in cesarean sections.

SECONDARY OUTCOMES:
Dose that achieves "adequate" uterine tone | 3 minutes
  Determining dose that achieves "adequate" uterine tone as defined by obstetricians on a qualitative numerical scale defined prior to the study (0 to 10 with 0 being inability of uterus to contract (i.e. uterine atony) to 10 being fully contracting uterus; "adequate" would be >5 on the scale)
Need for additional uterotonic agents | 3 minutes
  Quantifying need for additional uterotonic agents as outlined by the postpartum hemorrhage guidelines set forth by ACOG
Frequency of side effects of methylergonovine | 30 minutes
  Determining frequency of side effects of methylergonovine, including blood pressure changes, especially if elevated >20% preoperative level), headache, nausea, and vomiting
Need for vasopressors | 3 minutes
  To determine if the patient requires a vasopressor (including phenylephrine, ephedrine, epinephrine, norepinephrine or vasopressin)?
Estimated blood loss | 2 hours
  Utilizing estimated blood loss by suction canister + estimated weight of blood on surgical lap
Computed blood loss | 2 hours
  Calculating changes in hematocrit (Hct preop - Hct postop)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Lindeman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided